CLINICAL TRIAL: NCT05365425
Title: Effect of Choline Fenofibrate on Carotid Atherosclerosis Estimated by 3D Ultrasound in Patients With Type 2 Diabetes and Combined Dyslipidemia
Brief Title: Choline Fenofibrate and Carotid Atherosclerosis in Patients With Type 2 Diabetes and Combined Dyslipidemia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-2111-720-003
Record Dates: First submitted 2022-03-16; First posted 2022-05-09 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Dyslipidemia; Atherosclerosis; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Dyslipidemias; Atherosclerosis; Diabetes Mellitus, Type 2 | interventions — policosanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tgfenon (Experimental): Choline fenofibrate (135mg as fenofibric acid) 1 tablet once daily oral administration regardless of diet
  Interventions: Drug: Choline fenofibrate
- Policosanol 10 (Active Comparator): Policosanol 10mg 1 tablet once daily oral administration
  Interventions: Drug: Policosanol

INTERVENTIONS:
Drug: Choline fenofibrate — choline fenofibrate 178.8mg (135mg as fenofibric acid)
  Other Names: Tgfenon
  Arms: Tgfenon
Drug: Policosanol — policosanol 10mg
  Other Names: Policosanol 10
  Arms: Policosanol 10

SUMMARY:
This is a randomized controlled study to assess the effect of choline fenofibrate compared with policosanol in Korean T2DM patients with asymptomatic atherosclerosis.

DETAILED DESCRIPTION:
In patients with type 2 diabetes with atherosclerotic combined dyslipidemia, the effect of choline fenofibrate on the progression of carotid intima media thickness and carotid artery plaque will be evaluated by 3D carotid ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes under treatment with HbA1c 6.0-10.0% at screening visit
* Male or female of 20 years or over
* Mixed dyslipidemia: triglyceride 200~499 mg/dL, HDL-cholesterol male ≤45 mg/dL or female ≤50 mg/dL
* Identified carotid artery plaque: carotid intima-media thickness (cIMT) ≥ 1.0 mm
* Creatinine ≤1.8 mg/dL

Exclusion Criteria:

* Dyslipidemia which requires other therapy: triglyceride ≥500 mg/dL or LDL-cholesterol ≥190 mg/dL
* Uncontrolled hypertension
* Severe renal dysfunction
* GOT/GPT >120/120 or chronic liver disease
* Pregnant or childbearing woman who does not have enough contraception
* Changes of medication related to chronic diseases (diabetes, hypertension, dyslipidemia, etc.) within 3 months
* Other antiplatlet medication such as cilostazol, clopidogrel (except aspirin)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Carotid intima media thickness | 24 week
  Maximum carotid IMT (mm)

SECONDARY OUTCOMES:
Area of carotid artery plaque | 24 week
  measured by ultrasound
Plaque characteristics | 24 week
  changes of non-calcified plaque volume (mm3)
Glucose homeostasis | 24 week
  changes of HbA1c (%)
Lipid metabolism | 24 week
  TG concentration, HDL-cholesterol concentration
Bioelectrical Impedance Analysis | 24 week
  Body composition of fat mass (kg)
Proteinuria | 24 week
  albumin-to-creatinine ratio (mg/g)
changes of gut microbiota | 24 week
  measured by 16S rRNA or metagenome sequencing, comparing the composition or each phylum/genus/species

CONTACTS AND LOCATIONS:
Locations (1):
- SNUBH, Seongnam-si, Gyeonggi-do, South Korea